CLINICAL TRIAL: NCT00716729
Title: Development of Outcome-measures for Physically Active Patients With Hip and Groin Pain
Status: Completed | Type: Observational
Sponsor: Amager Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Physiotherapist Kristian Thorborg, Amager Hospital
Other Study IDs: H-C-2007-0129
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2008-07

CONDITIONS: Hip Disability; Groin Disability
Keywords: Questionnaire; Hip; Groin; Disability; Strength; To develop two new outcome measures for patients with hip and groin disability

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pateints with longstanding hip and/groin pain

SUMMARY:
The aim of this study is to develop an evaluative questionnaire, to evaluate patients with hip and groin disability, and a strength measurement for the hip, for patients with hip and groin disability.

Both measurement instrument are aimed for evaluating the natural course and different treatment modalities in patients with hip and groin disability.

ELIGIBILITY:
Inclusion Criteria:

* Hip and/groin pain more than 6 weeks
* Physically active

Exclusion Criteria:

* Systemic diseases
* Physically inactive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hip and/groin pain for more than 8 weeks
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Patient reported questionnaire | 1-2 years

SECONDARY OUTCOMES:
Strength measurement for the hip | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Amager Hospital, Copenhagen, Copenhagen S, Denmark

REFERENCES:
- [Derived] Thorborg K, Holmich P, Christensen R, Petersen J, Roos EM. The Copenhagen Hip and Groin Outcome Score (HAGOS): development and validation according to the COSMIN checklist. Br J Sports Med. 2011 May;45(6):478-91. doi: 10.1136/bjsm.2010.080937. PMID 21478502